CLINICAL TRIAL: NCT04126083
Title: Lofexidine for Rapid Pre-Operative Opioid Tapering in Adults Undergoing Lumbar Spine Surgery
Brief Title: Lofexidine for Adults Undergoing Lumbar Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: USWM, LLC (dba US WorldMeds) (Industry)
Responsible Party: Principal Investigator, W. Michael Hooten, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0002763
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-01

CONDITIONS: Opioid Withdrawal
Keywords: Opioid tapering; Spine surgery
MeSH Terms: interventions — lofexidine

STUDY DESIGN:
Intervention Model Description: Open label design
Masking Description: Open label design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lofexidine (Experimental): Patients will receive lofexidine 0.54 mg 4 times daily and the baseline opioid dose will be reduced by 10% daily.
  Interventions: Drug: Lofexidine Oral Tablet

INTERVENTIONS:
Drug: Lofexidine Oral Tablet — lofexidine 0.54 mg 4 times daily

SUMMARY:
The primary objective is to investigate the effects of lofexidine in adults undergoing opioid tapering prior to elective lumbar spine surgery.

DETAILED DESCRIPTION:
In this clinical trial, an open label design will be used to facilitate opioid tapering during a 12-day period prior to elective spine surgery. The primary outcome measure of this study is the number of patients who achieve a 50% reduction in daily opioid dose at day 12.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years.
2. Chronic lumbar spine pain for ≥ 3 months duration.
3. Scheduled for elective lumbar spine surgery.
4. Daily morphine equivalent dose between 50 mg and 200 mg.

Exclusion Criteria:

1. Cancer-related pain.
2. Medical or surgical conditions that could be adversely impacted by opioid tapering or use of lofexidine including, but not exclusively limited to, cardiac disease, inflammatory bowel disease, renal or hepatic impairment, vascular disease, and history of anaphylaxis. Patients may be excluded for other comorbid medical or surgical conditions based on the physician investigator's discretion.
3. History of schizophrenia or other chronic psychiatric disorder that could be adversely impacted by opioid tapering or use of lofexidine. Patients may be excluded for other comorbid mental health conditions based on the physician investigator's discretion.
4. Neurological condition that impair functioning in an ambulatory setting or could be adversely impacted by opioid tapering or use of lofexidine including, but not exclusively limited to, Parkinson's disease, amyotrophic lateral sclerosis, or a dementing illness. Patients may be excluded for other neurological conditions based on the physician investigator's discretion.
5. Active substance abuse disorder.
6. Inability to function in an ambulatory care setting due to severe deconditioning requiring use of supportive gait aids including a cane or walker. Patients may be excluded for other functional problems based on the physician investigator's discretion.
7. History of adverse effects attributed to opioid tapering or lofexidine use.
8. Use of medications from drug classes known to have adverse interactions with lofexidine including, but not exclusively limited to, beta-blockers, calcium channel blockers, alpha 1 and 2 receptor antagonists, tricyclic antidepressants, benzodiazepines, and selective serotonin reuptake inhibitors. Patients may be excluded for use of other medications based on the physician investigator's and research pharmacy's discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M Hooten, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data plan is undetermined.

REFERENCES:
- [Background] Fishman M, Tirado C, Alam D, Gullo K, Clinch T, Gorodetzky CW; CLEEN-SLATE Team. Safety and Efficacy of Lofexidine for Medically Managed Opioid Withdrawal: A Randomized Controlled Clinical Trial. J Addict Med. 2019 May/Jun;13(3):169-176. doi: 10.1097/ADM.0000000000000474. PMID 30531234
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Lofexidine: Patients received lofexidine 0.54 mg 4 times daily and the baseline opioid dose was reduced by 10% daily.
  Lofexidine Oral Tablet: lofexidine 0.54 mg 4 times daily
Period: Overall Study
Arm/Group | Lofexidine
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lofexidine
Number analyzed (Participants) | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [40 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Opioid Tapering
Description: The number of patients who achieve a 50% reduction in daily opioid dose at day 12.
Time Frame: 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lofexidine
Number analyzed (Participants) | 6
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 12 days.
Arm/Group | Lofexidine
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lofexidine (N=6)
Orthostatic Hypotension (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT04126083/Prot_SAP_000.pdf